CLINICAL TRIAL: NCT07404345
Title: Efficacy of Low-Dose Apixaban Added to Standard Heparin Lock to Prevent Dysfunction of Tunneled Hemodialysis Catheters: A Randomized, PROBE, Parallel-Grupo Trial.
Brief Title: Low-Dose Apixaban Added to Standard Heparin Lock Versus Heparin Lock Alone to Prevent Tunneled Hemodialysis Catheters Dysfunction (APICATH-HD)
Acronym: APICATH-HD
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Civil de Guadalajara (Other)
Responsible Party: Principal Investigator, Juan Alberto Gomez Fregoso, Principal Investigator, Hospital Civil de Guadalajara
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: APICATH-HD-01
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Hemodialysis Access Failure; Kidney Disease, End-Stage; Hemodialysis Catheter
Keywords: Hemodialysis; Tunneled central venous catheter; Catheter dysfunction; Catheter Failure; Catheter thrombosis; Apixaban; Heparin lock; End-stage kidney disease; Vascular access; Anticoagulation; PROBE trial
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — apixaban; Vascular Access Devices

STUDY DESIGN:
Intervention Model Description: Participants are individually randomized in a 1:1 ratio to one of two parallel groups and remain in the assigned group throughout follow-up (no crossover). Randomization is generated a priori using permuted blocks with concealed allocation. Follow-up is conducted at each hemodialysis session, with administrative censoring at 24 months or earlier upon permanent catheter removal/exchange, loss of catheter function requiring definitive intervention, kidney transplant, modality change, withdrawal, or death. The trial uses a PROBE approach: open-label clinical management with blinded endpoint adjudication by an independent committee.
Masking Description: This is a randomized, open-label, parallel-group trial. Participants and treating clinicians are aware of treatment allocation, as no placebo is used. To minimize assessment bias, all primary and secondary outcomes related to catheter dysfunction and catheter-related infections are adjudicated by an independent committee blinded to treatment allocation. Data provided to the adjudication committee are de-identified and coded to conceal group assignment. This approach is consistent with a PROBE (Prospective, Randomized, Open-label, Blinded Endpoint) study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Heparin sodium lock solution (Active Comparator): Standard catheter care including intraluminal heparin lock per unit protocol.
  Interventions: Drug: Heparin sodium lock solution
- Apixaban + Heparin Lock (Experimental): Standard catheter care plus apixaban 2.5 mg orally every 12 hours; same heparin lock protocol as control.
  Interventions: Drug: Apixaban + Heparin Lock

INTERVENTIONS:
Drug: Apixaban + Heparin Lock — Heparin sodium catheter lock solution (1,000 IU/mL) instilled into each lumen of the tunneled hemodialysis catheter at the end of each dialysis session, using a volume equal to the catheter manufacturer's priming volume per lumen. Plus Apixaban 2.5 mg orally every 12 hours, started after randomization and continued until administrative censoring at 24 months or earlier study end (e.g., catheter removal/exchange, modality change, kidney transplant, withdrawal, or death). Dose interruptions, bleeding events, and adherence are recorded per protocol.
  Arms: Apixaban + Heparin Lock
Drug: Heparin sodium lock solution — Heparin sodium catheter lock solution (1,000 IU/mL) instilled into each lumen of the tunneled hemodialysis catheter at the end of each dialysis session, using a volume equal to the catheter manufacturer's priming volume per lumen. The same lock protocol is used in both study arms.
  Arms: Heparin sodium lock solution

SUMMARY:
This randomized, single-center, PROBE trial evaluates whether adding low-dose apixaban (2.5 mg orally every 12 hours) to standard intraluminal heparin lock prolongs primary functional patency of tunneled hemodialysis catheters compared with standard heparin lock alone. Adult patients on hemodialysis with a recently implanted, functioning tunneled catheter (≥8 days) will be randomized 1:1 and followed up to 24 months (or until catheter loss). Primary outcome is time to first intervention for catheter dysfunction or definitive catheter loss. Secondary outcomes include primary-assisted and secondary patency, thrombotic dysfunction, rescue procedures, catheter-related infection, bleeding (ISTH), and mortality. Outcomes adjudication will be blinded.

DETAILED DESCRIPTION:
Design: Single-center, randomized (1:1), parallel-group, superiority trial with a PROBE strategy (open-label clinical management; blinded outcome adjudication by an independent committee).

Arms / Interventions Arm 1: Control - Heparin Lock Alone

Intervention Name:

Heparin Lock

Description:

Intraluminal heparin lock after each hemodialysis session as standard care. Heparin concentration is 1,000 IU/mL, with per-lumen volume equal to the priming volume specified by the catheter manufacturer.

Arm 2: Intervention - Apixaban Plus Heparin Lock

Intervention Name:

Apixaban

Description:

Intraluminal heparin lock identical to the control arm (standard care; heparin 1,000 IU/mL with per-lumen volume according to device priming volume), plus systemic anticoagulation with apixaban 2.5 mg orally every 12 hours.

Population: Adults (≥18 years) on hemodialysis with a tunneled double-lumen catheter (Palindrome®) in the internal jugular (right/left) or femoral (right/left) position, functioning and ≥8 days post-implantation, without early dysfunction.

Procedures: Per dialysis session, record prescribed/achieved blood flow, inline pressures, alarms, recirculation, line inversion, and lock details; document formal interventions for dysfunction (rt-PA instillation, related angioplasty, over-the-wire exchange), and evaluate infections using CDC criteria.

Follow-up: Each dialysis session and monthly safety/adherence checks; administrative censoring at 24 months or upon catheter loss/replacement, refractory infection, switch to AV access, transplant, death, or end of study.

Safety: Bleeding surveillance (ISTH). Temporary interruption rules for procedures/bleeding/concomitant drugs. Independent DSMB with one interim analysis at ~50% of primary events using O'Brien-Fleming boundaries.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years with end-stage kidney disease (CKD stage 5) receiving maintenance hemodialysis or initiating hemodialysis.
* Recently placed tunneled, double-lumen central venous hemodialysis catheter (tunneled CVC) in place for ≥8 days, with a post-placement radiograph confirming adequate tip position.
* Permitted catheter insertion sites: right internal jugular, left internal jugular, right femoral, or left femoral vein.
* Adequate initial catheter function, defined as ability to achieve the prescribed extracorporeal blood flow (suggested ≥300 mL/min) for ≥8 days after catheter placement.
* Conventional in-center hemodialysis schedule (2-3 sessions/week) at the study unit, with expected ability to complete follow-up for up to 24 months.
* Written informed consent provided.
* Willingness to receive only the protocol-assigned antithrombotic prophylaxis and to avoid non-study systemic anticoagulants or antiplatelet agents during the study period.

Exclusion Criteria:

* Non-tunneled hemodialysis catheter, subclavian catheter, or intracaval catheter placement not consistent with the protocol (e.g., catheter located in the SVC/IVC without a subcutaneous tunnel, or catheter location/site not permitted by the study).
* Tunneled catheter placed <8 days before randomization or radiographically confirmed catheter tip malposition at screening.
* Active bleeding; active peptic ulcer disease; or clinically significant gastrointestinal bleeding within the past 30 days; uncorrectable INR >1.5; platelet count <100,000/µL.
* High bleeding risk (HAS-BLED score >3) or major bleeding that is active or recent.
* Known coagulopathy; history of heparin-induced thrombocytopenia (HIT); or allergy/hypersensitivity to heparin, citrate, or rt-PA (alteplase).
* Severe hepatic impairment (e.g., Child-Pugh class C), clinically significant liver dysfunction that contraindicates DOAC therapy, or ongoing hemodialysis with regional citrate anticoagulation that cannot be modified per protocol.
* Active catheter exit-site infection or bloodstream infection/bacteremia at the time of randomization.
* Concomitant use of other systemic anticoagulants (e.g., warfarin, low-molecular-weight heparin, other DOACs) or high-intensity antiplatelet therapy (e.g., dual antiplatelet therapy).
* Pregnancy or breastfeeding.
* Women of childbearing potential who are unwilling to use a highly effective contraception method during the study and for 48 hours after the last dose of study medication.
* Life expectancy <6 months, current palliative/hospice care, or planned kidney transplant within ≤3 months.
* Concurrent participation in another clinical trial that could interfere with the study interventions or outcomes.
* Venography demonstrating significant venous stenosis involving the superior vena cava (SVC) or inferior vena cava (IVC).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Clinically significant catheter dysfunction | From randomization (T0) up to 24 months
  Time from randomization to the first clinically significant catheter dysfunction event, defined as either: (1) use of intraluminal thrombolytic therapy (alteplase/rt-PA), or (2) definitive catheter loss (permanent catheter removal or over-the-wire exchange) due to catheter dysfunction. The following are not considered events for the primary outcome: line reversal, flushing with crystalloid, postural changes, or radiography with subsequent manipulation unless they are followed by thrombolytic use or definitive catheter loss.

SECONDARY OUTCOMES:
Minor catheter dysfunction requiring simple maneuvers. | From randomization (T0) up to 24 months
  Time from randomization to the first episode of catheter dysfunction managed with simple maneuvers only, defined as any of the following performed to restore adequate dialysis without thrombolytic therapy or catheter exchange: line reversal, flushing/permeabilization with crystalloid, patient repositioning, or radiography followed by catheter manipulation/repositioning. Episodes that subsequently require alteplase/rt-PA or definitive catheter loss are counted as primary outcome events (and are not classified as 'minor').
Rescue procedures for catheter dysfunction (number of procedures per participant) | Up to 24 months
  Total number of protocol-defined rescue procedures performed for catheter dysfunction per participant during follow-up (line reversal, flushing/permeabilization with crystalloid, patient repositioning, or radiography followed by catheter manipulation/repositioning)
Catheter-related infection rate (per 1,000 catheter-days) | Up to 24 months
  Rate of catheter-related infection events defined using CDC criteria, expressed as events per 1,000 catheter-days during follow-up. Catheter-days are calculated from randomization until catheter removal/exchange or censoring.
Major bleeding (ISTH) | Up to 24 months
  Occurrence of major bleeding events defined according to ISTH criteria during follow-up.
Clinically relevant non-major bleeding (ISTH) | Up to 24 months
  Occurrence of clinically relevant non-major bleeding events defined according to ISTH criteria during follow-up.
All-cause mortality | Up to 24 months
  Death from any cause during follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Juan A Gomez Fregoso, Nephrologist, Principal Investigator — Antiguo Hospital Civil de Guadalajara "Fray Antonio Alcalde" (Servicio de Nefrología)
Locations (1):
- Antiguo Hospital Civil de Guadalajara "Fray Antonio Alcalde", Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the results reported in publications will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 6 months after primary publication and ending 5 years thereafter
Access Criteria: Requests will be reviewed by the study steering committee. Data will be shared with qualified researchers for methodologically sound proposals, after approval and execution of a data use agreement. Only de-identified data will be provided; no direct identifiers will be shared